CLINICAL TRIAL: NCT00752557
Title: A PHASE 2, MULTICENTER, RANDOMIZED, ACTIVE-CONTROLLED, PARALLEL-GROUP, DOSE-FINDING AND SAFETY STUDY OF RECOMBINANT HUMAN BONE MORPHOGENETIC PROTEIN-2 (RHBMP-2)/CALCIUM PHOSPHATE MATRIX(CPM) IN SUBJECTS WITH DECREASED BONE MINERAL DENSITY
Brief Title: Study Evaluating Changes In Bone Mineral Density (BMD), And Safety Of Rhbmp-2/CPM In Subjects With Decreased BMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3100N0-2213; B1921002 (Other: Alias Study Number); 2007-007456-34 (EudraCT Number)
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis
Keywords: Bone mineral density; bone morphogenetic protein; osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Diphosphonates; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): rhBMP-2/CPM , 1.0 mg/mL
  Interventions: Drug: rhBMP-2/CPM injection and bisphosphonates, calcium, and vitamin D (oral bisphosphonate therapy)
- 2 (Experimental): rhBMP-2/CPM , 2.0 mg/mL
  Interventions: Drug: rhBMP-2/CPM injection and bisphosphonates, calcium, and vitamin D (oral bisphosphonate therapy)
- 3 (Active Comparator): Oral bisphosphonate therapy (standard of care)
  Interventions: Drug: bisphosphonates, calcium, and vitamin D

INTERVENTIONS:
Drug: rhBMP-2/CPM injection and bisphosphonates, calcium, and vitamin D (oral bisphosphonate therapy) — Single, unilateral intraosseous injection of 6mL of rhBMP-2/CPM , 1.0 mg/mL.
  Arms: 1
Drug: rhBMP-2/CPM injection and bisphosphonates, calcium, and vitamin D (oral bisphosphonate therapy) — Single, unilateral intraosseous injection of 6mL of rhBMP-2/CPM , 2.0 mg/mL.
  Arms: 2
Drug: bisphosphonates, calcium, and vitamin D — Oral bisphosphonate therapy
  Arms: 3

SUMMARY:
The main purpose of this study is to assess whether a locally-administered rhBMP-2/CPM injection can rapidly increase bone mass in subjects at high risk for osteoporotic fractures of the hip. All subjects will receive standard treatment for low bone mass, consisting of bisphosphonates, calcium, and vitamin D (all taken by mouth). Subjects that are randomly selected to receive treatment with rhBMP-2 will receive an injection directly into the hip. The injection is given in a surgery room using a light anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling, ambulatory (with or without assistive device), postmenopausal females, age greater than 65 years.
* BMD T-score (total hip or femoral neck) of -2.5 or less in at least 1 hip. Subjects with BMD T-scores of -2.0 or less may be enrolled if at least one of the following risk factors is also present:
* Age greater than 75 years
* Family (maternal) history of fragility fracture
* Previous fragility fracture (self) after age 45
* Subjects may either be treatment naïve or on a previously-established regimen ( greater than 1year, but less than 5 years duration) of bisphosphonate therapy. Subjects must be willing to comply with 1of the 3 protocol-designated oral bisphosphonates (risedronate, alendronate, or ibandronate sodium) with risedronate considered as first-line therapy.

Exclusion Criteria:

* Metabolic bone disorder or disease affecting bone and mineral metabolism (eg, Paget's disease, vitamin D deficiency [ less than 20 ng/mL], hyperparathyroidism, renal osteodystrophy, osteomalacia, hypocalcemia, hypercalcemia).
* Coagulopathy and/or history of venous thromboembolic events (deep vein thrombosis, pulmonary embolus, retinal vein thrombosis) within the past 12 months.
* Inflammatory arthritis including rheumatoid, psoriatic, or crystal-induced (gouty) arthritis, or those associated with systemic lupus erythematosus (SLE), spondyloarthropathy, Reiters syndrome, or Crohns disease.

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (28):
  - Arizona Research Center, Inc., Phoenix, Arizona
  - John C. Lincoln Hospital - Deer Valley, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - UC Davis Medical Center, Sacramento, California
  - Florida Hospital Deland, DeLand, Florida
  - Florida Orthopaedic Associates, P.A., DeLand, Florida
  - Florida Research Associates, LLC, DeLand, Florida
  - Victoria Park Imaging, DeLand, Florida
  - Diagnostic Professionals, Inc., Fort Lauderdale, Florida
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - Suncoast Clinical Research Inc, New Port Richey, Florida
  - Coastal orthopedic and Sports Medicine, New Port Richey, Florida
  - Westside Regional Medical Center, Plantation, Florida
  - Florida Arthritis & Osteoporosis Center, Port Richey, Florida
  - Medical Center of Trinity, Trinity, Florida
  - Intensive Research Unit, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - Creighton University Osteoporosis Research Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Prairie Lakes Healthcare Systems, Watertown, South Dakota
  - Brown Clinic, Watertown, South Dakota
  - Cool Spring Interventional, PLLC, Franklin, Tennessee
  - Center for Women's Health Research at Meharry Medical College, Nashville, Tennessee
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Andre Dumont Ziekenhuis - ZOL, Campus Andre Dumont, Waterschei (Genk)
- Poland (3):
  - Synexus Polska Sp. z o.o., Warsaw, Masovian Voivodeship
  - Radiologica, Pracownia Rezonansu Magnetycznego i Tomografii Komputerowej, Warsaw, Masovian Voivodeship
  - Centralny Szpital Kliniczny MSWiA, Zaklad Diagnostyki Radiologicznej, Warsaw, Masovian Voivodeship
- Spain (2):
  - Clinica Ruber, Madrid
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3100N0-2213&StudyName=Study%20Evaluating%20Changes%20In%20Bone%20Mineral%20Density%20%28BMD%29%2C%20And%20Safety%20Of%20Rhbmp-2/CPM%20In%20Subjects%20With%20Decreased%20BMD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 centers in the United States of America, Belgium, and Poland.
Pre-assignment Details: Treatment assignments were stratified by previous osteoporosis (OP) therapy regardless of rhBMP-2/CPM treatment assignment; bisphosphonate, calcium, vitamin D were provided to all participants as background concomitant OP therapy.
Groups:
- Standard of Care Control: Participants had received systemic osteoporosis therapy with an oral bisphosphonate plus supplemental calcium, and vitamin D as prescribed by the study physician.
- rhBMP-2/CPM 1.0 mg/mL: Participants had received 1 mg/mL rhBMP 2/CPM administered via intraosseous injection administered percutaneously to the proximal femur. Participants in treatment groups additionally received SOC treatment for OP.
- rhBMP-2/CPM 2.0mg/mL: Participants had received 2 mg/mL rhBMP 2/CPM administered via intraosseous injection administered percutaneously to the proximal femur. Participants in both injected treatment groups additionally received SOC treatment for OP.
Period: Overall Study
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPM 2.0mg/mL
Started | 17 | 16 | 17
Completed | 12 | 11 | 11
Not Completed | 5 | 5 | 6
Not completed — Withdrawal by Subject | 4 | 3 | 3
Not completed — Unspecified resaons | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The as-treated population included randomly assigned participants who received at least 1 dose of rhBMP-2/CPM or comparator agent. Participants in the as-treated population are grouped according to the treatment they received (not the treatment to which they were randomly assigned).
Groups:
- rhBMP-2/CPm 2.0 mg/mL: Participants had received 2 mg/mL rhBMP 2/CPM administered via intraosseous injection administered percutaneously to the proximal femur. Participants in treatment groups additionally received SOC treatment for OP.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL | Total
Number analyzed (Participants) | 17 | 15 | 14 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.35 (5.454) | 75.93 (5.271) | 73.21 (5.041) | 74.15 (5.304)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 14 | 46
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) Measured by Dual-Energy X-ray Absorptiometry (DXA)
Description: Evaluating local changes (expected increases) in BMD after administration of rhBMP-2/CPM, compared to those observed with systemic osteoporosis therapy alone. Alternatively, if changes in the total area surrounding the proximal femur are observed, bone mineral content (BMC) may instead be applied for the primary measure. BMD is defined as a derived measure of bone density, generated by dividing the bone mineral content value obtained from a bone densitometry technique (for example, DXA) by the total area of the region scanned.
Time Frame: Baseline, 12 months post dose
Population: As-treated population included randomly assigned participants who received at least 1 dose of rhBMP-2/CPM or comparator agent. Participants were grouped as per the treatment they received (not to the treatment they were randomly assigned). Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: gram per centimeter squared (g/cm^2)
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 14 | 12 | 14
gram per centimeter squared (g/cm^2)
  Total hip | -0.0026 (0.018) | 0.1299 (0.045) | 0.1196 (0.063)
  Intertrochanter | -0.0029 (0.020) | 0.1063 (0.066) | 0.1192 (0.063)
  Trochanter | -0.0091 (0.023) | 0.1197 (0.066) | 0.0869 (0.073)
  Femoral neck | 0.0058 (0.021) | 0.2408 (0.111) | 0.2120 (0.117)

2. Primary Outcome: Time Course Distribution of Volumetric BMD for the Hip Under Study (HUS) for Total Hip
Description: Time course distribution of volumetric Bone mineral density (BMD) for hip is assessed by volumetric Quantitative Computed Tomography (vQCT) technique which is a 4-detector spiral (helical) computed tomography (CT) scanner with designated calibration phantom, obtain a CT scan of the proximal femora (bilateral simultaneous acquisition with volumetric rendering) to identify the specified region of interests (ROIs) for volumetric parameter to be quantified, reconstruct images of both hips and send reconstructed data (in electronic format). The vQCT regions of interest are cortical, the subcortical and trabecular. Cortical and the subcortical BMD are distinguished from trabecular effects. Peeled trabecular BMD reflects the subtraction of the extended CPM. Integral BMD reflects the cortical, subcortical, and peeled trabecular regions (minus the extended Calcium phosphate matrix [CPM]).
Time Frame: At Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram per centimeter cubed (mg/cm^3)
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 13 | 11 | 14
milligram per centimeter cubed (mg/cm^3)
  Cortical + Sub-Cortical | 136.8 (16.91) | 165.6 (18.37) | 151.6 (26.07)
  Peeled Trabecular | 45.1 (16.02) | 77.8 (23.07) | 88.4 (37.63)
  Integral | 181.9 (20.60) | 243.4 (31.04) | 240.0 (45.31)

3. Secondary Outcome: Summary of Volumetric Density of Cortical and Trabecular Bone Calculated by Quantitative Computed Tomography (vQTC)
Description: Here, measurement of density of cortical and trabecular bone in various regions of interest (ROIs) in the femoral neck, proximal shaft, and individual trochanters and was calculated by Quantitative Computed Tomography (vQTC) in ROIs.
Time Frame: 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 5 | 7 | 6
mg/cm^3
  Cortical Bone | 2.5782 (0.16805) | 2.4259 (0.24267) | 2.5128 (0.17484)
  Trabecular Bone | 0 (0) | 4.7073 (2.40500) | 4.2205 (1.63904)

4. Secondary Outcome: Number Participant Responses to Injectability Questionnaire Injected Population
Description: Investigator documents preparation of the study medication evaluates injectability and product placement relative to desired location (for participants in active treatment groups). Surgeon performing the injection had to complete the questionnaire that evaluates ease of preparing the study medication, ability to administer study medication, and ability for the study medication to remain in the location it was administered.
Time Frame: Participants were monitored after treatment administration (dosing period)
Population: Only those participants who were injected with rhBMP-2/CPM were included in the injected population. Any participant who received SOC alone was excluded from this population.
Measure: Number; unit: Participants
Arm/Group | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 15 | 14
Participants
  Ease of Preparing-satisfactory | 15 | 14
  Ease of Preparing-unsatisfactory | 0 | 0
  Ease of Injecting-satisfactory | 15 | 11
  Ease of Injecting-unsatisfactory | 0 | 3
  Ability to inject entire volume- satisfactory | 13 | 12
  Ability to inject entire volume- unsatisfactory | 2 | 2
  Localization within Proximal Femur-satisfactory | 15 | 11
  Localization within Proximal Femur-unsatisfactory | 0 | 2
  Missing | 0 | 1

5. Secondary Outcome: Number of Participants With Any Significant Changes in Serum Biomarkers of Bone Turnover From Baseline
Description: Participants with significant change in serum biomarkers of bone formation and resorption from baseline are reported. Significant changes were judged by investigator.
Time Frame: Baseline up to 12 months
Population: As-treated population included randomly assigned participants who received at least 1 dose of rhBMP-2/CPM or comparator agent. Participants in the as-treated population are grouped according to the treatment they received (not the treatment to which they were randomly assigned).
Measure: Number; unit: participants
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 17 | 15 | 14
participants | 0 | 0 | 0

6. Primary Outcome: Timecourse Distribution of Volumetric Bone Mineral Density (BMD) for the Hip Under Study (HUS). Volume of Interest: Femoral Neck
Description: Evaluating local changes (expected increases) in BMD after administration of rhBMP-2/CPM, compared to those observed with systemic osteoporosis therapy alone. Alternatively, if changes in the total area surrounding the proximal femur are observed, bone mineral content (BMC) may instead be applied for the primary measure.
Time Frame: At Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 13 | 11 | 14
mg/cm^3
  Cortical +Sub Cortical | 144.3 (16.81) | 166.3 (31.06) | 164.4 (29.37)
  Peeled Trabecular | 61.1 (14.39) | 165.0 (59.13) | 159.3 (38.97)
  Integral | 205.4 (23.02) | 331.3 (73.99) | 323.7 (58.96)

7. Secondary Outcome: Percentage Change From Baseline in Areal Bone Mineral Density (BMD) for Contralateral Total Hip
Description: Evaluating local changes (expected increases) in BMD after administration of rhBMP-2/CPM, compared to those observed with systemic osteoporosis therapy alone. The percentage change from baseline in BMD for total hip (assessed by DXA) is presented for the contralateral (untreated) hip below.
Time Frame: 36 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Number analyzed (Participants) | 10 | 12 | 12
Percent change | 0.73 (0.057) | 0.71 (0.045) | 0.71 (0.110)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of written informed consent through 3 years, month 36 (Visit 10) for SOC participants and through Visit 12 (month 60) for participants who either received 1.0 mg/mL or 2.0 mg/mL of rhBMP-2/CPM.
Description: The as-treated population included randomly assigned participants who received at least 1 dose of rhBMP-2/CPM or comparator agent. Participants in the as-treated population are grouped according to the treatment they received (not the treatment to which they were randomly assigned).
Arm/Group | Standard of Care Control | rhBMP-2/CPM 1.0 mg/mL | rhBMP-2/CPm 2.0 mg/mL
Serious Adverse Events (participants affected / at risk) | 3/17 | 7/15 | 7/14
Other Adverse Events (participants affected / at risk) | 13/17 | 15/15 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Control (N=17) | rhBMP-2/CPM 1.0 mg/mL (N=15) | rhBMP-2/CPm 2.0 mg/mL (N=14)
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Control (N=17) | rhBMP-2/CPM 1.0 mg/mL (N=15) | rhBMP-2/CPm 2.0 mg/mL (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymph node calcification (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Chronotropic incompetence (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Choroidal haemorrhage (Eye disorders) | 1 | 0 | 0
Dark circles under eyes (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Macular generation (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
retinal haemorrhage (Eye disorders) | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 6 | 5
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 3
Breakthrough pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Gait deviation (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 1
Injection site discharge (General disorders) | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 2 | 0
Injection site mass (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 5
Injection site swelling (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 2 | 1
Peripheral swelling (General disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 2
Soft tissue inflammation (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 2
Coccidioidomycosis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 5 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Chest X-ray abnormal (Investigations) | 0 | 1 | 0
Scan bone marrow abnormal (Investigations) | 0 | 1 | 0
Urine output increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Iodine deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 12 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aortic calcification (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0
Vascular calcification (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
46 participants enrolled; further enrollment suspended due to safety signal. Participants completed long-term follow up per protocol; extra 2 years per protocol amendment. Sample size small to draw conclusions, to conduct efficacy interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study participating sites. Investigator may not disclose previously undisclosed confidential other than study results.